CLINICAL TRIAL: NCT01985399
Title: Neurocognitive Effects and Tolerability of Efavirenz in Aging HIV-infected Individuals ("SHAC Neuro Study")
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Principal Investigator, Philip Grant, Principle Investigator, Stanford University
Other Study IDs: SHAC Neuro Study
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: HIV; AIDS
Keywords: HIV; AIDS; Aging
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EFV containing ARV regimen: Pts on Efavirenz containing ARV regimen will have neuropsychological testing performed
  Interventions: Behavioral: Neuropsychological testing
- Non -EFV ontaning ARV regimen: Pts on a Non-Efavirenz containing ARVregimen will have neuropsychological testing measures performed
  Interventions: Behavioral: Neuropsychological testing

INTERVENTIONS:
Behavioral: Neuropsychological testing — Neuropsychological testing

SUMMARY:
Investigators hypothesize that older HIV-infected individuals (i.e., >50 years old) on efavirenz (EFV)-containing antiretroviral therapy (ART) will have significantly worse neurocognitive function than older individuals on non-EFV-containing ART.

DETAILED DESCRIPTION:
With the aging of the HIV-infected population in the United States and elsewhere, neurocognitive dysfunction will likely become an increasingly common problem. Older individuals could be at increased risk for efavirenz-associated adverse effects due to impaired metabolism, increased drug-drug interactions, and lower physiologic reserve, but there are few data on the long-term safety of efavirenz (and other antiretrovirals) in older individuals with HIV.

The Stanford HIV Aging Cohort (SHAC) is an ideal setting to study potential neurologic effects of antiretrovirals in aging patients. SHAC is an ongoing longitudinal study initiated in 2008 to evaluate aging in virologically-suppressed HIV-infected individuals. The cohort is supported through multiple grants including a grant from the State of California's HIV Research Program as well as a NIH supplemental grant. As of September 2013, approximately 150 virologically-suppressed HIV-infected adults have been enrolled. In addition to enrolling patients with good adherence to ART, the cohort purposefully excludes subjects with active substance abuse, unstable medical conditions, and psychiatric illnesses to limit potential confounding the study end points. Recently, an NIH supplemental grant (AI069556) was received which will expand the SHAC to 300 HIV-infected subjects. The median age of the subjects in the cohort is in the mid-50's allowing an ample number of older subjects for our planned studies.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment into SHAC (Stanford HIV Aging cohort)
* Age over 50 years of age
* Stable antiretroviral therapy containing EFV- or PI-containing ART (but not both) for at least 6 months
* HIV RNA levels of <200 copies/mL for at least 6 months excluding blips (i.e., a single measurement between 200-500 copies/mL preceded and followed by measurements of <200 copies/mL) while on ART.

Exclusion Criteria:

* Completed treatment for any acute systemic infection (other than HIV-1) less than four weeks before study entry
* Any active brain infection (except for HIV-1), brain neoplasm, or space-occupying brain lesion.
* Any active psychiatric illness including schizophrenia, severe depression, or severe bipolar affective disorder that, in the opinion of the investigator, could confound the analysis of the neuropsychological test results.
* Active drug or alcohol abuse that, in the investigator's opinion, could prevent compliance with study procedures or confound the analysis of study endpoints.
* Hospitalization within 30 days of study entry
* Receipt of systemic chemotherapy within 30 days of study entry
* Unable to provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 individuals on an EFV-containing regimen and 50 individuals on a protease-inhibitor (PI)-containing regimen
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Compare a composite measure of neurocognitive function in older individuals on EFV-containing ART vs. non-EFV-containing ART. | one year
  Neurocognitive function will be assessed using a detailed battery of neuropsychologic tests including timed gait, grooved pegboard with the dominant and non-dominant hands, the Rey auditory verbal learning test trials I-VII, trail making parts A and B, Rey auditory verbal learning test trial VIII 30-min delay, controlled oral word association test and paced auditory serial addition task. This battery has been used extensively in previous studies in HIV. Z-scores for each neurocognitive test, based on age-adjusted norms, and a composite Z-score will be calculated. The Z-score represents the amount, in standard deviation units, that the subject's test result deviates from population means.
  In addition to neurocognitive function, the level of depression and anxiety and sleep quality will be evaluated using validated instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Grant, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University AIDS Clinical Trials Unit, Palo Alto, California, United States